CLINICAL TRIAL: NCT00740402
Title: Motor Learning of a Planning Task in Stroke Patients
Brief Title: Motor Learning of a Planning Task in Stroke Patients: the Maze Paradigm Measured Through Time and Error as Variables
Status: Completed | Type: Observational
Sponsor: Faculdades Metropolitanas Unidas (Other)
Responsible Party: Acquisition of manual motor hability in patients after stroke, Camila Torriani
Other Study IDs: GPalma; GPalma 123 (Other: UNICID/USP)
Record Dates: First submitted 2008-08-22; First posted 2008-08-25 (Estimated); Last update posted 2010-04-16 (Estimated); Status verified 2008-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — no biospecimens are to be retained
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to investigate the process of acquiring a motor skill subject in post-stroke, comparing them with healthy subjects.

DETAILED DESCRIPTION:
20 post-stroke patients were comprised to the experimental group (EG) and 20 health subjects were included to the control group (CG. Inclusion criteria: chronic stroke, single stroke event, lesion in anterior circulation, right handed subjects, MEEM over 23 points. The task consisted in a maze paradigm, made by pencil and paper, with the non affected side for EG and left upper extremity for CG. The instruction was given to the subjects to complete the task as fast as possible. The study consisted in three phases: acquisition (AQ)with 30 trials, transfer (TR, short retention (R1)and long term retention (R2 both with 5 trials.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 65
* Injury in territory of movement earlier, as shown by examination of image and finding medical neurologist
* Time of injury over 6 months
* Single vascular event
* Right handed, by applying the Inventory of Dominance Side of Edinburgh Mini mental with scores over 23 points

Exclusion Criteria:

* Aphasia of understanding
* Instability clinic
* Other neurological diseases associated (Parkinson's disease, dementias, Alzheimer)

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients after stroke
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-01; Primary Completion 2008-07 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
TIME | 3 times in a week (acquisition, transfer an retention phase)
  time (in seconds)

SECONDARY OUTCOMES:
error | 3 times in a week (acquisition, transfer an retention phase)
  number of mistakes made by the subjects

CONTACTS AND LOCATIONS:
Overall Officials: Camila Torriani, doctor, Study Chair — University of Sao Paulo
Locations (1):
- University Center of Metropolitan United, São Paulo, São Paulo, Brazil